CLINICAL TRIAL: NCT02218554
Title: Performance Evaluation of the Micromedic BRONJ Risk Assessment in Vitro Diagnostic Assay.
Acronym: BRONJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Micromedic Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-BNJ-001-PR
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-05

CONDITIONS: Bisphosphonate-related Osteonecrosis of the Jaw
Keywords: BRONJ
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Subject has been diagnosed with BRONJ
  Interventions: Genetic: BRONJ
- Control Group (No Intervention): Subject has not developed any signs or symptoms of BRONJ

INTERVENTIONS:
Genetic: BRONJ — collection of the blood sample from the subject for evaluation of the Micromedic BRONJ Risk Assessment in vitro Diagnostic Assay
  Arms: Study Group

SUMMARY:
To evaluate the performance of the Micromedic BRONJ Risk Assessment in vitro assay (the "BRONJ Assay") in identifying Multiple Myeloma (MM) and/or other cancer subjects at risk for developing Bisphosphonate-related Osteonecrosis of the Jaw (BRONJ) following intravenous (IV) administration of Bisphosphonates (BP).

DETAILED DESCRIPTION:
The Micromedic BRONJ Assay is intended for the qualitative analysis of genetic changes which may be indicative of increased risk to develop BRONJ osteonecrosis of the jaw (ONJ) following IV administration of drugs of the Bisphosphonate family.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Study Group (all of the following):

1. Subject is ≥18 years old
2. Subject is or was a Multiple Myeloma and/or other cancer patient who is or has been IV treated with the BP zoledronic acid and/or pamidronate disodium; Or; Subject is or was a Multiple Myeloma and/or other cancer patient who is or has been IV treated with the BP zoledronic acid and/or pamidronate disodium and was also treated by oral BP such as sodium alendronate, and in the opinion of the PI, IV treatment was significant enough to be considered as the cause for BRONJ
3. Subject has been diagnosed with BRONJ at stages 1 or 2 or 3 according to AAOMS (American Association of Oral and Maxillofacial Surgeons)
4. Subject has signed the informed consent or consent can be waived

Inclusion Criteria Control Group (all of the following):

1. Subject is ≥18 years old
2. Subject is or was a Multiple Myeloma and/or other cancer patient who is, or has been IV treated with the BP zoledronic acid and/or pamidronate disodium for at least two (2) years (continuously or cumulatively)
3. Subject has not developed any signs or symptoms of BRONJ
4. Subject has signed the informed consent or consent can be waived

Exclusion Criteria:

1. Subject has been treated with irradiation to the jaws or head and neck at levels exceeding 35 Gy
2. Pregnant or lactating women
3. Subject has been treated with either bevacizumab or sunitimib
4. Subject has been treated with Allogeneic hematopoietic stem cell transplantation (HSCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
For each subject, the primary endpoint is the presence or absence of SNPs or other genetic alterations obtained from the assay for blood samples | up to 2 years

SECONDARY OUTCOMES:
For each subject, the secondary endpoint is the presence or absence of additional/alternative SNPs or other genetic alterations using GWAS analysis and/or Full Exome Sequencing (FES) from the assay for blood samples | up to 2 years

OTHER OUTCOMES:
Safety endpoints will include adverse events (AEs), including serious AEs (SAEs) whether or not deemed related to study procedures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noam Yarom, Dr., Principal Investigator — Sheba MC
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel